CLINICAL TRIAL: NCT00035828
Title: A Blinded Study Comparing the Safety and Efficacy of a Fully Human Anti-IL8 Monoclonal Antibody (ABX-IL8) to Placebo in Patients With Chronic Bronchitis and COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abgenix (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABX-0209
Record Dates: First submitted 2002-05-06; First posted 2002-05-07 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic
Keywords: COPD; Chronic bronchitis; Chronic obstructive pulmonary disease; Shortness of breath; Dyspnea; Bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Dyspnea; Bronchitis | interventions — ABX-Interleukin 8

INTERVENTIONS:
Drug: ABX-IL8

SUMMARY:
To determine if ABX-IL8 will improve shortness of breath.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is defined as a disease state characterized by the presence of airflow obstruction due to chronic bronchitis or emphysema. The airflow obstruction is generally progressive, may be accompanied by airway hyper-reactivity, and may be partially reversible. Inflammation in the lungs is triggered by exposure to inhaled toxic substances that can lead to tissue damage, mucous secretion, airways narrowing and tissue destruction.

Interleukin-8 (IL-8) plays a major role in elevating sputum in patients with COPD and may contribute to tissue destruction. Therefore, the highly specific antibody to IL-8 (such as ABX-IL8) may help to reduce mucous production and tissue destruction.

ELIGIBILITY:
Inclusion Criteria:

* > 50 years old
* > 20 pack-year of smoking
* Diagnosed with COPD and chronic bronchitis

Exclusion Criteria:

* Patients with bronchiectasis, cystic fibrosis, tuberculosis, asthma, alpha-1 antitrypsin deficiency, CHF
* Require oxygen therapy
* Uncontrolled hypertension
* HIV or Hepatitis
* Recent history of COPD exacerbation
* Patients with cancer
* Recent history of infection

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2001-12; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Locations (1):
- Abgenix, Fremont, California, United States